CLINICAL TRIAL: NCT04524936
Title: Relation of Serum Irisin Levels, Non-Alcoholic Fatty Liver Disease, Glucose and Lipid Metabolism Parameters in Obese Children
Brief Title: Serum Irisin Levels in Obese Children
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, gökçen ulualan, Principal Investigator, Eskisehir Osmangazi University
Other Study IDs: I-OBESITY
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Serum Irisin Levels in Obese Children
Keywords: irisin; obesity; children; non-alcoholic fatty liver disease
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- obese patient with non-alcoholic fatty liver disease
  Interventions: Diagnostic Test: blood sample
- obese patient without non-alcoholic fatty liver disease
  Interventions: Diagnostic Test: blood sample
- control group
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample

SUMMARY:
Irisin is a myokine induced by exercise, that converts white fat tissue to brown fat tissue, thereby increases thermogenesis and energy expenditure. The aim of this study is to determine the relationships between serum irisin levels and glucose and lipid parameters in obese children with and without non-alcoholic fatty liver disease (NAFLD). A total of 60 pubertal obese children (age range: 11-18 years) will be included in the study. 30 of these patients will be had NAFLD. The control group consisted of 28 healthy children who will be similar in age and sex to the obese group.

DETAILED DESCRIPTION:
Obesity and related complications (non-alcoholic fatty liver disease (NAFLD), type 2 diabetes mellitus (DM)) have become an important public health problem. Their prevalence continues to increase worldwide in children. Therefore, estimating potential biomarkers that can cause obesity and related complications can be important in their treatment.

Irisin, a myokine, first described by Boström et al. (5) in 2012, is released into the circulation as a product of Fibronectin type III domain-containing 5 (FNDC5) gene activated by increased expression of peroxisome proliferator-activated receptor-ɣ coactivator-1' (PGC1)-α in the muscle cell along with exercise. The circulating irisin increases the expression of UCP1 mRNA in WAT cells. As a result, WAT cells are converted into BAT cells. Thus, irisin is involved in termogenesis and energy consumption.

Conflicting results have been reported in studies investigating the relationship between irisin level and obesity and related complications. Irisin was thought to play a role in the development of obesity. It has been suggested that it may be an alternative treatment agent for obesity and glucose tolerance. In some studies, irisin levels were found to be higher in obese children and adults than in healthy controls, low in some, and not different in others.

There is limited data in the relevant literature about the relationships between childhood obesity and irisin, as well as between NAFLD and irisin. In our study, we aimed to determine whether serum irisin levels are related to anthropometric measurements and metabolic and biochemical parameters in obese children with and without NAFLD.

Sixty obese pubertal patients (31 girls, 29 boys), aged between 11-18 years, admitted to the pediatric endocrinology outpatient clinic of our hospital wiil be included in the study. These patients will be divided into two groups with and without NAFLD. Patients with another disease or any drug use will be not included in the study. The control group consisted of 28 healthy children (14 girls, 14 boys) who will be similar in age and sex to the obese group.

Physical examination will be done in all children. Body weight (BW) and height will be measured. Body mass index (BMI) values will be compared with BMI curves according to age and gender. BMI≥95.p will be considered as obese. Subcutaneous fat thickness will be measured from the triceps and biceps regions by using a caliper. Waist circumference will be measured in the horizontal plane midway between lowest rib and the iliac crest. Hip circumference will be measured over the widest area of the hips. Waist-to-hip ratio will be calculated.

After one night fasting, two venous serum samples will be taken for irisin levels and biochemical analysis. Glucose, total cholesterol (TC), triglycerides (TG), low density lipoprotein-cholesterol (LDL-C), high density lipoprotein-cholesterol (HDL-C), ALT, AST, GGT levels, insulin levels will be determined.

Venous serum samples for the irisin levels will be stored at -80°C until the analysis. Serum irisin levels will be measured.

The homeostasis model assessment of insulin resistance (HOMA-IR) will be calculated using the following formula: fasting insulin level (uIU/ml) x fasting glucose (mg/dl) / 405. A HOMA-IR value >5.22 in males and >3.82 in females will be considered having IR.

Hepatobiliary ultrasound (US) will performed for NAFLD

ELIGIBILITY:
Inclusion Criteria:

* BMI≥95.p
* Puberty
* The control group will be similar in age and sex to the obese group.

Exclusion Criteria:

* viral hepatitis,
* autoimmune hepatitis,
* primary sclerosing cholangitis,
* hemochromatosis,
* drug-induced liver disease,
* Wilson disease,
* α-1 antitrypsin deficiency,
* type 1 DM,
* pancreatitis,
* thyroid disease,
* renal failure,
* estrogen, progesterone, glucocorticoids, insulin, UDCA, iron, interferon, antibiotics, levothyroxine sodium, metformin, antiepileptic drug used

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pubertal children
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
serum irisin levels | 1 day
  Serum irisin levels were measured and compared in three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University Faculty of Medicine, Eskişehir, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No